CLINICAL TRIAL: NCT05051709
Title: Can Hypermobility of First Ray Affect Surgical Treatment of Hallux Valgus: Randomized Control Trial
Brief Title: Can Hypermobility of First Ray Affect Surgical Treatment of Hallux Valgus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hawler Medical University (Other)
Responsible Party: Principal Investigator, Sherwan Ahmed Ali Hamawandi, Assistant professor of orthopedic surgery, Hawler Medical University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: HMU/Sherwan12
Record Dates: First submitted 2021-09-11; First posted 2021-09-21 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Hallux Valgus
Keywords: Hallux valgus; First ray hypermobility; Fusion; Corrective osteotomy; Functional outcome
MeSH Terms: conditions — Hallux Valgus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Foot with no fusion (Active Comparator)
  Interventions: Procedure: Corrective osteotomy
- Foot with fusion (Active Comparator)
  Interventions: Procedure: Fusion of First ray

INTERVENTIONS:
Procedure: Corrective osteotomy — First metatarsal distal corrective osteotomy
  Arms: Foot with no fusion
Procedure: Fusion of First ray — Fusion of first ray with soft tissue procedure
  Arms: Foot with fusion

SUMMARY:
Hallux valgus can be associated with hypermobility of 1st ray. Surgical decision for hallux valgus can be affected by hyper mobility of 1st ray so our clinical trial involved patients with bilateral hallux valgus were planned to underwent fusion of 1st ray and soft tissue correction plus bonionectomy for one foot and for other foot surgical treatment involves corrective osteotomy and soft tissue procedure plus bonionectomy without fusion of 1st tarsometatarsal joint.

ELIGIBILITY:
Inclusion Criteria:

* Hallux Valgus with 1st ray hypermobility

Exclusion Criteria:

1. Generalized Ligament laxity
2. Previous foot and ankle surgery
3. Diabetes Mellitus

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-09-15 (Estimated); Primary Completion 2022-09-15 (Estimated); Study Completion 2023-09-15 (Estimated)

PRIMARY OUTCOMES:
American foot and ankle score | This score was assessed one year after surgery
  American foot and ankle score involved 9 section
Foot and Ankle Disability Index | This score was assessed one year after surgery
  Foot and Ankle Disability Index involved 26 sections

CONTACTS AND LOCATIONS:
Locations (1):
- Hawler Medica University, Erbil, Iraq

IPD SHARING:
Plan to Share IPD: Undecided
Later we will decide